CLINICAL TRIAL: NCT00275301
Title: Brain Correlates of Olanzapine Treatment Response in BPD
Brief Title: PET Imaging and Olanzapine Treatment in Borderline Personality Disorder
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Minnesota (Other)
Collaborators: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0506M70791
Record Dates: First submitted 2006-01-10; First posted 2006-01-11 (Estimated); Results first posted 2017-05-23 (Actual); Last update posted 2017-05-23 (Actual); Status verified 2017-04

CONDITIONS: Borderline Personality Disorder
Keywords: Borderline Personality Disorder; BPD; PET; olanzapine; brain
MeSH Terms: conditions — Borderline Personality Disorder | interventions — Olanzapine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Open-label Olanzapine. (Experimental): Open-label Olanzapine.
  Interventions: Drug: olanzapine

INTERVENTIONS:
Drug: olanzapine — Olanzapine 2.5mg by mouth at bedtime x2 weeks, then Olanzapine 5mg by mouth at bedtime x2 weeks, then Olanzapine 7.5mg by mouth at bedtime x4 weeks.
  Other Names: Zyprexa

SUMMARY:
The overall design of the study is to perform both a PET and MRI scan on objectively identified borderline personality disorder patients, to treat them with olanzapine for 8 weeks, and to then re-scan the patients with PET.

DETAILED DESCRIPTION:
The primary objective of this proposed study will be to compare the baseline PET scan to the endpoint scan in 15 BPD patients who have been treated with olanzapine. The comparison of the scans will be done through a statistical image analysis, using a pixel-by-pixel group mean subtraction strategy with appropriate correction for multiple comparisons. In an exploratory fashion we will compare frontal and temporal regions of interest to address hypotheses of which areas of the brain might show changes with olanzapine treatment.

A secondary objective is to use a normal database to compare the baseline PET scan of the 15 patients in a medication free state to normal subjects. The advantage of this strategy is the ability to closely match subjects by gender and age. As noted earlier, Dr. Pardo has data on 35 control subjects studied on the same scanner we plan to use for this study.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-45 years
2. Diagnosis: borderline personality disorder by DSM-IV criteria
3. Gender: Female
4. May have history of substance use and other Axis II disorders

Exclusion Criteria:

1. Axis I diagnosis of schizophrenia, schizoaffective disorder, or bipolar I disorder during the subject's lifetime. No current major depression or PTSD.
2. Treatment with psychotropic medication in the previous month.
3. Medical disorder that would influence outcome of the study - e.g. epilepsy, thyroid disease, HIV, etc.
4. Medical disorder that would not allow use of olanzapine
5. Active substance abuse or dependence
6. Previous adverse reaction to olanzapine
7. Females whom are pregnant or nursing

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 19 (Actual)
Dates: Start 2005-12; Primary Completion 2008-04 (Actual); Study Completion 2008-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: S. Charles Schulz, MD, Principal Investigator — University of Minnesota
Locations (1):
- University of Minnesota, Dept of Psychiatry, Minneapolis, Minnesota, United States

REFERENCES:
- See also: Treatment and Research Advancements Nat'l Assn for BPD — http://www.tara4bpd.org/bpd.html

RESULTS

PARTICIPANT FLOW:
Recruitment Details: All subjects were symptomatic volunteers from the community.
Pre-assignment Details: 19 subjects were enrolled. 5 early withdrawals. 14 subjects completed the entire study.
Groups:
- All Subjects Took Open-label Olanzapine.: All subjects took open-label olanzapine. Subjects tritrated to up to 10mg
Period: Overall Study
Arm/Group | All Subjects Took Open-label Olanzapine.
Started | 19
Completed | 14
Not Completed | 5
Not completed — Adverse Event | 5

BASELINE CHARACTERISTICS:
Population: 19 subjects were enrolled.
Groups:
- All Subjects Were Open-label and Took the Same Dose.: This was an open-label study so all subjects were in the same group.
Arm/Group | All Subjects Were Open-label and Took the Same Dose.
Number analyzed (Participants) | 19
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 19
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 26.4 (7.56)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14
  Male | 5
Region of Enrollment [Number; unit: participants]
  United States | 19

OUTCOME MEASURES:

1. Primary Outcome: Change in Brain Metabolism From Baseline to Eight Weeks as Seen in PET Scan
Description: The primary aim of this imaging study was to examine the effect of olanzapine on brain metabolism over the eight weeks of administration. To compare the baseline PET scan to the endpoint scan,
Time Frame: Baseline to 8 weeks
Measure: Mean (Standard Deviation); unit: Standard uptake value
Arm/Group | All Subjects Were Open-label and Took the Same Dose.
Number analyzed (Participants) | 19
Standard uptake value | 11.5 (.5)
Statistical Analysis 1: Comparison: All Subjects Were Open-label and Took the Same Dose; Examination of relationship between Borderline Personality Disorder symptoms and brain metabolism at baseline; Test type: Superiority or Other; p < 0.05, Regression, Linear

ADVERSE EVENTS:
Time Frame: 8 weeks
Description: All subjects took open-label olanzapine.
Arm/Group | All Subjects Were Open-label and Took the Same Dose.
Serious Adverse Events (participants affected / at risk) | 0/14
Other Adverse Events (participants affected / at risk) | 14/14
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | All Subjects Were Open-label and Took the Same Dose. (N=14)
Sedation (Nervous system disorders) | 14 (20) — All 14 subjects reported sedation.

LIMITATIONS AND CAVEATS:
Small number of subjects (14) analyzed. 19 subjects were enrolled but 5 subjects withdrew early from the study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No